CLINICAL TRIAL: NCT03993028
Title: The Effects of Sex, Body Mass Index, Day-to-Day Subject Variability and Variability of a Single Device When Volume-Averaged Thoracic Bioconductance is Measured With the ProLung Test
Brief Title: The Effects of Sex, Body Mass Index, Day-to-Day Subject Variability for the ProLung Test and Variability of a Single Device When Volume-Averaged Thoracic Bioconductance is Measured With the ProLung Test
Status: Completed | Type: Observational
Sponsor: Fresh Medical Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: PL-209
Record Dates: First submitted 2015-11-25; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the repeatability of the ProLung Test

DETAILED DESCRIPTION:
This repeatability study of the ProLung Test enrolled sixty subjects, 30 male and 30 female, half of each sex with a body mass index (BMI) of 30 or more, and half with a BMI of 28 or less. Each subject was scanned twice on Day One and twice on Day Two. All scans were done by the same operator on the same device. Fifty-nine subjects produced evaluable data. Four models (algorithms) were tested.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 70 years
* Able to understand and fulfill all requirements of this protocol
* Provide signed informed consent

Exclusion Criteria:

* Pacemaker or other implanted medical device
* Current life-threatening medical condition
* Current or recent use of systemic corticosteroids
* Pregnant or lactating
* Unusually strenuous exercise within previous 24 hours
* Current abuse of alcohol or drugs
* Medical or anatomical condition that precludes testing of all 62 measurement points
* Other condition or reason at the discretion of the Principal Investigator or medical monitor

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Quantify EPN Scanner variability in transcutaneous volume-averaged thoracic bio-conductance when measured twice on the same subjects by the same operator on a single same day using the same EPN Scanner | 1 day
  The null hypothesis is that same-day variability has no effect on scan results (i.e. when scanned twice on the same day).
Quantify day-to-day within-subject variability when the same operator uses the same EPN Scanner on the same subjects to measure transcutaneous volume-averaged thoracic bio-conductance on two different days within one week. | 1 week
  The null hypothesis is that day-to-day variability has no effect on scan results (i.e. when scanned twice on separate days).
Effects of BMI and Sex on transcutaneous volume-averaged thoracic bio-conductance | 1 week
  The null hypothesis is that BMI has no effect on scan results. The null hypothesis is that sex has no effect on scan results.
Number of participants with device-related adverse events from thoracic bio-conductance measurement. | 1 day
  time to complete scan.